CLINICAL TRIAL: NCT00832377
Title: Prospective, Open-label, Single-arm Study to Evaluate Efficacy and Safety of Combination Therapy of Timolol and Dorzolamide (COSOPT) as Initial Treatment for Patients With Normal Tension Glaucoma
Brief Title: COSOPT (Timolol/Dorzolamide Combination) Normal Tension Glaucoma Study (MK0507A-161)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0507A-161; 2009_524
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Timolol/Dorzolamide (Experimental): Timolol/Dorzolamide, 1 drop, twice daily, for 12 weeks
  Interventions: Drug: timolol/dorzolamide combination

INTERVENTIONS:
Drug: timolol/dorzolamide combination — Timolol/Dorzolamide, 1 drop, twice daily, for 12 weeks
  Other Names: Cosopt

SUMMARY:
A study to evaluate the effect of the 12-week treatment with timolol/dorzolamide combination eyedrops (COSOPT) on decrease in intraocular pressure (IOP) at 2 hours after the study drug administration

ELIGIBILITY:
Inclusion Criteria:

* Patients who have not been treated with a glaucoma medication within 6 weeks prior to study participation after diagnosis with primary open-angle glaucoma
* Patients with primary open-angle glaucoma based on gonioscopy
* Patients with normal tension glaucoma diagnosed based on accompanying optic disc cupping and reappearance of visual field defect corresponding to retinal nerve fiber layer defect.
* Subjects with < 22 mm Hg of diurnal IOP measured using Goldmann applanation tonometer (every two hours between 9 a.m. and 5 p.m.)

Exclusion Criteria:

* Patients with another type of glaucoma but primary open-angle glaucoma
* Patients treated with other glaucoma medications within 6 weeks prior to study participation
* Patients with a history of chronic ocular inflammation or recurrent ocular inflammation
* Patients using contact lenses
* Patients who are allergic to timolol or dorzolamide
* Patients with a history of any of the following COSOPT (timolol/dorzolamide combination) contraindications:

  * Reactive airway diseases
  * Sinus bradycardia, second or third degree atrioventricular block, overt cardiac failure, cardiogenic shock
  * Severe renal impairment
* Patients with a history of significant ocular trauma or intraocular surgery within 6 months before participating the study, or intraocular laser surgery within 3 months before the participating the study
* Patients with a history of a corneal disease
* Patients who are using steroid or used the drug for more than 2 weeks within 12 months before participating the study
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2010-03-12 (Actual); Study Completion 2010-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kim TW, Kim M, Lee EJ, Jeoung JW, Park KH. Intraocular pressure-lowering efficacy of dorzolamide/timolol fixed combination in normal-tension glaucoma. J Glaucoma. 2014 Jun-Jul;23(5):329-32. doi: 10.1097/IJG.0b013e3182741f4d. PMID 23377586

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 participants were actually screened. Among them, 7 participants failed in screening (2 participants withdrew and 5 did not meet eligibility criteria). Therefore 37 participants were considered to have enrolled.
Period: Overall Study
Arm/Group | Timolol/Dorzolamide
Started | 37
Completed | 36
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Timolol/Dorzolamide
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Peak Intraocular Pressure (IOP) Measured Two Hours After Study Drug Administration at Week 12 Compared to Baseline IOP.
Description: The therapeutic goal of normal tension glaucoma treatment includes lowering IOP to prevent progression of damage in optic nerves or vision. In this trial, IOP was measured with the same tonometer throughout the study. A decreased IOP from baseline is considered an improvement.
  IOP was measured in both eyes and the eye with the higher IOP was used for the participant.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol/Dorzolamide
Number analyzed (Participants) | 36
mmHg | -3.73 (2.28)
Statistical Analysis 1: Comparison: Timolol/Dorzolamide; Test type: Superiority or Other; p < 0.0001, paired t-test — Week 12 peak IOP vs. baseline

2. Secondary Outcome: Mean Change in Trough IOP Measured Right Before Study Drug Administration at Week 12 Compared to Baseline IOP.
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol/Dorzolamide
Number analyzed (Participants) | 36
mmHg | -3.22 (2.14)
Statistical Analysis 1: Comparison: Timolol/Dorzolamide; Test type: Superiority or Other; p < 0.0001, paired t-test — Week 12 trough IOP vs. baseline

3. Secondary Outcome: Mean Change in IOP 8 Hours After the Study Drug Administration at Week 12 Compared to Baseline IOP
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol/Dorzolamide
Number analyzed (Participants) | 36
mmHg | -3.78 (2.40)
Statistical Analysis 1: Comparison: Timolol/Dorzolamide; Test type: Superiority or Other; p < 0.0001, paired t-test — Week 12 8-HR IOP vs. baseline

4. Other Pre Specified Outcome: Baseline IOP
Description: Baseline IOP was measured at ~9 AM of first day of treatment period.
  IOP was measured in both eyes and the eye with the higher IOP was used for the participant.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol/Dorzolamide
Number analyzed (Participants) | 36
mmHg | 15.60 (2.46)

ADVERSE EVENTS:
Arm/Group | Timolol/Dorzolamide
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 24/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Timolol/Dorzolamide (N=37)
Eye irritation (Eye disorders) | 22 (32)
Ocular hyperaemia (Eye disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.